CLINICAL TRIAL: NCT02122042
Title: Hyperbaric Oxygen Therapy Can Improve Cognitive Deficits Post Low Grade Glioma Removal Surgery - Randomized Prospective Trial
Brief Title: Hyperbaric Oxygen Therapy Can Improve Cognitive Deficits Post Low Grade Glioma Removal Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Shai Efrati, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 64/14
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Post Low Grade Glioma Surgery; Cognitive Deficits
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBOT (Experimental): Group will be treated with HBOT for 60 treatments in 3 months.
  Interventions: Biological: HBOT
- Control/Crossover (Other): Control for 3 months without treatment, and then HBOT for 60 treatments in 3 months.
  Interventions: Biological: HBOT

INTERVENTIONS:
Biological: HBOT
  Other Names: HBOT of 2 ATA for 90 minutes O2 100%, for 60 treatments

SUMMARY:
The aim of the current study is to evaluate, in a prospective cross-over, randomized study, the effect of hyperbaric oxygen therapy (HBOT) on patients with chronic impairment after low grade glioma tumor removal surgery

ELIGIBILITY:
Inclusion Criteria:

* Post low grade glioma (WHO I-II) removal surgery 3-12 months prior to the inclusion in the study.
* All patients have to have persistent cognitive impairment (Mindstream score should be at least one SD lower than average) regarding without noticeable improvement during the last month prior to their enrolment.
* Age 18 years or older.

Exclusion Criteria:

* Dynamic neurologic/cognitive improvement or worsening during the past month; Previous brain radiotherapy and/or radiosurgery. Steroids dependence Chemotherapy in the past month or scheduled in the next 3 months Seizures 1 month previous to inclusion Had been treated with HBOT for any other reason 1 month prior to inclusion; Have any other indication for HBOT; Chest pathology incompatible with pressure changes; Inner ear disease; Patients suffering from claustrophobia; Inability to sign written informed consent; Smoking patients will not be allowed to smoke during the study and if they would not comply with this demand they will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive functions | 6 months
  Cognitive function will be assessed using the one-hour Mindstreams Computerized Cognitive Test Battery at baseline, 3 months and 6 months to intervention.

SECONDARY OUTCOMES:
Quality of Life | 6 months
  Quality of live will be evaluated by the EQ-5D,SS-QOL ו SF36 , QLQ-BN20, questionnaires at baseline , 3 months and 6 months to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel, Israel